CLINICAL TRIAL: NCT05533814
Title: A Multicenter, Open-Label, Prospective Study With an Extension Phase to Evaluate the Efficacy and Safety of Perampanel Monotherapy in Untreated Subjects With Focal Onset Seizures With or Without Focal to Bilateral Tonic-Clonic Seizures
Brief Title: A Study to Evaluate the Efficacy and Safety of Perampanel Monotherapy in Untreated Participants With Focal Onset Seizures With or Without Focal to Bilateral Tonic-clonic Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-M082-606
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy
Keywords: Epilepsy; Focal onset seizures; Focal to bilateral tonic-clonic seizures; Fycompa; Seizures; Monotherapy; Open-label
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perampanel (Experimental): Participants will be administered oral perampanel at a starting dose of 2 milligram (mg) per day. Doses of perampanel will then be up titrated in increments of 2 mg every 2 weeks up to maximum of 8 mg per day at the discretion of the investigator, and the dose may be administered up to maximum tolerated dose (MTD) according to the clinical response and tolerance of individual participants.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel tablets.
  Other Names: Fycompa; E2007

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of perampanel monotherapy measured by the seizure-free rate during the Maintenance Period (24 weeks) of the Treatment Phase in untreated participants with focal onset seizures (FOS) with or without focal to bilateral tonic-clonic seizures (FBTCS).

DETAILED DESCRIPTION:
The study will consist of a Core Study (36 weeks) and an Extension Phase (24 weeks). Core Study will consist of 4 weeks Pre-treatment Phase or Baseline and 32 weeks Treatment Phase (8 weeks Titration period and 24 weeks Maintenance period).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, age 4 years or older
2. Diagnosis of epilepsy with FOS with or without FBTCS according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures (2017), established by clinical history and an electroencephalogram (EEG)
3. Newly diagnosed or recurrent epilepsy with at least 2 unprovoked seizures (excluding focal non-motor seizures) separated by a minimum of 24 hours in the 1 year before Visit 1 (baseline)

Exclusion Criteria:

1. Focal non-motor seizures only
2. Generalized epilepsies or seizures such as absences and/or myoclonic seizures, or Lennox Gastaut syndrome
3. History of status epilepticus within 1 year before Visit 1 (baseline)
4. History of psychogenic non-epileptic seizures within 5 years before Visit 1 (baseline)
5. Progressive central nervous system (CNS) disease (including degenerative CNS diseases, progressive tumors, and dementia), or clinically significant psychological or neurological disorders
6. History of suicidal ideation/attempt within 5 years before Visit 1 (baseline)
7. Evidence of clinically significant active hepatic disease, or other clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigators could affect the participant safety or interfere with the study assessments
8. History of any type of brain or central nervous system surgery within 1 year before Visit 1 (baseline)
9. Newly started ketogenic diet or has been on ketogenic diet for less than 5 weeks before Visit 1 (baseline)
10. Multiple drug allergies or a severe drug reaction to anti-epileptic drugs (AEDs), including dermatological (example, Stevens-Johnson syndrome), hematological, or organ toxicity reactions
11. Hypersensitive to perampanel or ingredients of this drug
12. Participant with genetic problems including galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
13. Use of intermittent rescue medication on 2 or more occasions within 4 weeks before Visit 1 (baseline)
14. History of receiving any AED (except for occasional use less than 2 weeks of AEDs as rescue treatment), antipsychotics, or anti-anxiety drugs within 12 weeks before Visit 1 (baseline)
15. History of receiving any AED (including rescue treatment) for more than 2 weeks in total within 2 years before Visit 1 (baseline)
16. Has received prior treatment with perampanel
17. Females of child bearing potential who are breastfeeding or pregnant at Visit 1 (baseline), or who do not consent to employ contraception
18. Currently enrolled in another clinical study or have used any investigational drug/biologics or device within 28 days or 5*half-life, whichever is longer
19. Participant who did not consent to having at least 2 weeks of washout period before Visit 2, if known to take Cytochrome P4503A (CYP3A) inducing drugs or foods on Visit 1 (including, but not limited to the following) - Carbamazepine, enzalutamide, mitotane, phenytoin, phenobarbital, amobarbital, secobarbital, rifabutin, rifampicin, food containing St. John's Wort (hypericum perforatum), bosentan, efavirenz, etravirine, modafinil, armodafinil, rufinamide, nevirapine, oxcarbazepine, and glucocorticoid (except for topical use)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Will Achieve Seizure Freedom During the 24-weeks Maintenance Period | Up to 24 weeks

SECONDARY OUTCOMES:
Percentage of Participants Who Will Achieve Seizure Freedom During the Total 48-weeks Treatment Period (24-weeks Maintenance Period Plus 24-weeks Extension Phase) | Up to 48 weeks
Percentage of Participants With at Least 50 Percent (%) and 75% Reduction in Seizure Frequency During the 24-weeks Maintenance Period | Up to 24 weeks
  50% responder rate is defined as the percentage of participants with greater than or equal to (>=) 50% reduction in seizure frequency. 75% responder rate is defined as the percentage of participants with >=75% reduction in seizure frequency.
Percentage of Participants With at Least 50% and 75% Reduction in Seizure Frequency During the 24-weeks Extension Phase | Up to 24 weeks
  50% responder rate is defined as the percentage of participants with >=50% reduction in seizure frequency. 75% responder rate is defined as the percentage of participants with >=75% reduction in seizure frequency.
Median Percent Change From Baseline in Partial Onset Seizure Frequency per 28 Days at the End of 8 Weeks Titration Period | Baseline up to Week 8 of Titration Period
Median Percent Change From Baseline in Partial Onset Seizure Frequency per 28 days at the End of 24 Weeks Maintenance Period | Baseline up to Week 24 of Maintenance Period
Median Percent Change From Baseline in Partial Onset Seizure Frequency per 28 days at the End of 24 Weeks Extension Phase | Baseline up to Week 24 of Extension Phase
Percentage of Participants Remaining on Perampanel Treatment at the end of Maintenance Period | Week 24 of Maintenance Period
  The retention rate is defined as the percentage of participants remaining on perampanel treatment at the end of Maintenance Period after initiating treatment.
Percentage of Participants Remaining on Perampanel Treatment at the end of Extension Phase | Week 24 of Extension Phase
  The retention rate is defined as the percentage of participants remaining on perampanel treatment at the end of Extension Phase after initiating treatment.
Number of Participants With One or More Treatment-emergent Adverse Events (TEAEs) | Up to 60 weeks
  A TEAE is defined as an adverse event (AE) that emerges during treatment, having been absent at pretreatment (Baseline) or reemerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous. An AE is defined as any untoward medical occurrence in a participant administered an investigational product. An AE does not necessarily have a causal relationship with a medicinal product.
Number of Participants With Abnormal Vital Sign Values | Up to 60 weeks
  Vital sign parameters will include diastolic and systolic blood pressure (BP), pulse rate, respiratory rate, body temperature and body weight.
Number of Participants With Clinically Significant Laboratory Values | Up to 60 weeks
  Laboratory parameters will include hematology and blood chemistry.

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Eisai Site #9, Cheongju-si
  - Eisai Site #4, Daegu
  - Eisai Site #8, Daegu
  - Eisai Site #3, Daejeon
  - Eisai Site #10, Jeonju
  - Eisai Site #1, Seoul
  - Eisai Site #2, Seoul
  - Eisai Site #5, Seoul
  - Eisai Site #6, Seoul
  - Eisai Site #7, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.